CLINICAL TRIAL: NCT07311369
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase Ⅱa Study to Evaluate the Safety and Efficacy of HL-1186 Tablets for Postoperative Pain Management in Abdominal Surgery
Brief Title: Evaluate the Safety and Efficacy of HL-1186 Tablet for Postoperative Pain Management in Abdominal Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Yidian Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Shanghai Huilun Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PY-HL-1186-AS-Ⅱa-01
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Moderate to Severe Acute Postoperative Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HL-1186 (Experimental): Participants will be randomized to either the HL-1186 group or placebo group, and administer study drug every 12 hours for 4 consecutive doses
  Interventions: Drug: HL-1186
- HL-1186 placebo (Placebo Comparator): Participants will be randomized to either the HL-1186 group or placebo group, and administer study drug every 12 hours for 4 consecutive doses
  Interventions: Drug: HL-1186 placebo

INTERVENTIONS:
Drug: HL-1186 — HL-1186 tablet for oral administration.
  Arms: HL-1186
Drug: HL-1186 placebo — HL-1186 placebo tablet for oral administration.
  Arms: HL-1186 placebo

SUMMARY:
This is a multiple-center, randomized, double-blind, placebo-controlled study design evaluating the safety, efficacy, and pharmacokinetics (PK) parameter of HL-1186 tablet for postoperative pain management in abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 75 years old, gender is not limited.
2. 18 kg/m2 ≤ Body Mass Index (BMI) ≤ 30kg/m2.
3. Scheduled to undergo abdominal surgeries under general anesthesia.
4. Able to understand the research process and the use of pain scales, and communicate effectively with researchers.

Exclusion Criteria:

1. Prior history of surgery at the same site, and this may affect pain perception at the surgical site per investigator's judgments.
2. Allergy to any component of the investigational product, to perioperative anesthetic/analgesic/antiemetic agents, or to ≥3 substance allergies.
3. Unstable angina, myocardial infarction, severe arrhythmias (e.g., third-degree atrioventricular block), New York Heart Association (NYHA) class III or higher cardiac function, recurrent asthma, etc., within screen period, and deemed ineligible per investigator's judgments.
4. High bleeding risk conditions: Congenital bleeding disorders (e.g., hemophilia), platelet function abnormalities (e.g., idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, congenital platelet function abnormalities), active bleeding, etc., and deemed ineligible per investigator's judgments.
5. For female participants: Pregnant or lactating (within 1 year postpartum).
6. Participants with childbearing potential planning conception/sperm/egg donation within 6 months post-treatment, or unwilling to use effective contraception (abstinence, barrier methods, oral contraceptives, intrauterine device, or sterilization).
7. Judgment by the investigator that the participant should not enter the study due to other conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
SPID48 | 0 to 48 hours
  SPID48: Time-weighted Sum of the Pain Intensity Difference (SPID) as recorded on an NRS (Numeric Rating Scale, 0 =no pain to 10 =worst possible pain) at rest 0 to 48 hours after the first dose of study drug. The score range was -480 (worst score) to 480 (best score).

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Day 1 to Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No